CLINICAL TRIAL: NCT04960046
Title: A Comparison Between a Paracoracoid Approach and a Costoclavicular Approach for the Placement of Infraclavicular Perineural Catheters in Hand Surgery: a Prospective Randomized Controlled Trial.
Brief Title: A Comparison Between a PC and a CC Approach for the Placement of Infraclavicular Perineural Catheters in Hand Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 21.114
Record Dates: First submitted 2021-07-02; First posted 2021-07-13 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Postoperative Pain; Anesthesia, Local
Keywords: Infraclavicular perineural catheters; Hand surgery
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Intervention Model Description: Single-center, prospective, randomized controlled, triple blind
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: Randomized, triple-blind controlled study (participant, surgeon and evaluator).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Infraclavicular nerve block using a costoclavicular approach (Active Comparator): The costoclavicular approach, more recently described, proposes an insertion of the needle under the lower edge of the clavicle but in a lateral way to the axillary artery which makes it possible to reach the nerves at a place where the 3 main nerve bundles are still joined together. The clustering of nerve structures at the injection site may facilitate the spread of local anesthetics.
  Interventions: Procedure: Placement of an infraclavicular perineural catheter using a costoclavicular approach
- Infraclavicular nerve block using a paracoracoid approach (Placebo Comparator): The paracoracoid approach involves inserting a needle under the lower rim of the clavicle below the coracoid process. This approach makes it possible to reach the 3 different nerve bundles, located around the axillary artery, which are involved in the sensitivity of the hand.
  Interventions: Procedure: Placement of an infraclavicular perineural catheter by paracoracoid approach

INTERVENTIONS:
Procedure: Placement of an infraclavicular perineural catheter using a costoclavicular approach — The high-frequency linear probe will be used to image the axillary artery in the long axis and nearby nerve structures of interest, namely the posterior, lateral and medial bundles. The plane chosen will be located inferior to the clavicle, also in its distal third. The needle will be inserted with a latero-medial orientation in the plane. The initial injection will be a single injection laterally to the axillary artery, where the three nerve bundles are still joined together.
  The catheter will then be positioned and its location verified by injecting an additional 5 mL of bupivacaine into the catheter under direct ultrasound visualization. Catheter fixation will be standardized to minimize the risk of accidental displacement and the point of entry of the catheter to the skin will be covered with an opaque dressing.
  Arms: Infraclavicular nerve block using a costoclavicular approach
Procedure: Placement of an infraclavicular perineural catheter by paracoracoid approach — The high-frequency linear probe will be used to image the axillary artery in the short axis and nearby nerve structures of interest, namely the posterior, lateral and medial bundles. The plane chosen will be located inferior to the clavicle, in its distal third. The needle will be inserted with a cranio-caudal orientation in the plane. The initial injection will be a single injection posterior to the axillary artery, the expected distribution being a "U" distribution around the artery.
  The catheter will then be positioned and its location verified by injecting an additional 5 mL of bupivacaine into the catheter under direct ultrasound visualization. Catheter fixation will be standardized to minimize the risk of accidental displacement and the point of entry of the catheter to the skin will be covered with an opaque dressing.
  Arms: Infraclavicular nerve block using a paracoracoid approach

SUMMARY:
In outpatient hand surgery, 40% of patients report moderate to severe pain within 24 hours of the operation. Effective pain management is therefore essential to ensure a comfortable and safe return home for the patient.

Loco-regional anesthesia is the optimal method of analgesia for complex hand surgery. It involves the injection of a local anesthetic (LA) near the nerves responsible for the sensitivity of the arm. Following a single injection of long-acting local anesthetic, the maximum duration of analgesia is limited to approximately 13 hours, with great variability between individuals. In order to provide pain relief over a longer period of time, placing catheters near nerves has become a routine practice at the CHUM.

Infraclavicular nerve block is one of the most widely used loco-regional anesthesia techniques for hand surgery. This block can be achieved either by paracoracoid (PC) or costoclavicular (CC) approach. Both approaches are currently used at the CHUM.

The PC approach involves inserting a needle under the lower rim of the clavicle below the coracoid process. This approach makes it possible to reach the 3 different nerve bundles, located around the axillary artery, which are involved in the sensitivity of the hand.

The CC approach, more recently described, proposes an insertion of the needle under the lower edge of the clavicle but in a lateral way to the axillary artery which makes it possible to reach the nerves at a place where the 3 main nerve bundles are still joined together. The clustering of nerve structures at the injection site may facilitate the spread of local anesthetics.

Recent studies have demonstrated that the CC approach requires a smaller volume compared to the PC approach to achieve perineural blockade. The effective dose 90 (ED90) for the CC approach was 19 mL while it is 31 mL for the PC approach. This is explained by the greater proximity between the three nerve bundles targeted in the CC approach and a lower prevalence of anatomical variations at this level.

However, studies on the subject are rare and do not allow conclusions to be drawn on the superiority of either approach.

DETAILED DESCRIPTION:
The aim of this study is to determine whether the costoclavicular approach (CC) provides a better sensory block 48 hours after catheter installation than the infraclavicular block performed by the paracoracoid approach (PC).

In the context of continuous perineural blocks performed on an outpatient basis, LAs are delivered after insertion of a catheter by a low flow elastomeric pump (maximum 5 mL/h). Considering that the nerve structures are closer to each other with the CC approach, the investigators hypothesize that with the same mode of administration, the efficacy of the continuous block at 48 h obtained by the CC approach will be greater than the block produced by the PC approach.

Methods

Patients scheduled to undergo an upper limb surgery requiring a continuous infraclavicular nerve block will be contacted by a member of the research team before surgery to receive information regarding the study and obtain informed consent.

After obtaining consent, participants will be randomly assigned to two groups:

Group A: Placement of an infraclavicular perineural catheter by paracoracoid approach; Group B: Placement of an infraclavicular perineural catheter using a costoclavicular approach.

Only the anesthesiologist performing the technique and his assistant will know the group to which the patient has been assigned. The blocks will be carried out in a standardized manner and in accordance with the establishment's procedures. After bringing the patient to the induction room and installing the recommended monitoring equipment, the anesthesiologist will administer an intravenous premedication. The patient will be installed in a supine position. After disinfecting the skin, the anesthesiologist will inject a small amount of local anesthetic to numb the skin in the area where the block will be performed and then locate the nerve bundles under ultrasound guidance using the approach to which the patient has been assigned (Group A or B). When the area has been located, the injection of a local anesthetic (bupivacaine) will be performed and the catheter installed and fixed. Multimodal analgesia will be used for postoperative pain relief including acetaminophen, non-steroidal anti-inflammatory drugs and hydromorphone as needed.

Thirty minutes after the catheter insertion, a sensory-motor assessment of the blocked territory will be performed. During surgery, the patient may be sedated or receive general anesthesia at the discretion of the anesthesiologist. The surgery will be performed according to the usual procedure.

In day-care surgery, a disposable elastomeric pump will be installed to ensure the perineural infusion of LA. The patient will receive the usual information about postoperative analgesia and the use of the pump. Follow-up details will be reviewed with the patient prior to discharge from hospital.

A follow-up teleconsultation will be made the day after surgery and two days after surgery. As part of these calls, the following items will be assessed: sensory level and motor function of the forearm, level of pain and opioid use, presence of side effects, quality of sleep and satisfaction towards the analgesic technique used.

All patients will benefit from a daily follow-up call by nurses from the Acute Pain Service (APS) for up to 72 hours. In the absence of adverse effects, catheters will be removed by patients 72 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years old
* American Society of Anesthesiologists' classification 1 to 3
* Patients undergoing elective ambulatory hand surgery requiring the use of continuous infraclavicular nerve block

Exclusion Criteria:

* Contraindication to a peripheral nerve block
* Refusal of the patient or inability to consent
* Inability to communicate with the healthcare team or the research team
* Lack of access to the Teams telehealth platform
* Inability to understand the items of the different questionnaires
* Inability to understand ambulatory catheter follow-up instructions
* Pregnancy
* Obesity Body Mass Index > 40
* Pre-existing neurological deficit in the operated upper limb
* Anatomical malformation not allowing one of the study blocks to be performed
* Condition preventing measurement of the primary outcome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2025-04-02 (Actual); Study Completion 2025-04-04 (Actual)

PRIMARY OUTCOMES:
Proportion of patients presenting at least a partial sensory block in the four main nervous territories of the forearm | 48 hours after surgery
  Proportion of patients presenting at least a partial sensory block in the four main nervous territories of the forearm (ulnar, median, radial and musculocutaneous) using the score described by Boivin et al. after the surgery.
  A score of 0 to 2 will be assigned for each dermatome (0 = normal feeling; 1 = reduced sensation compared to the contralateral side (hypoesthesia); 2 = no feeling (anesthesia)).

SECONDARY OUTCOMES:
Proportion of patients presenting a motor block score greater than or equal to 1 in the four main nervous territories of the forearm | 24 and 48 hours after surgery
  Proportion of patients presenting a motor block score greater than or equal to 1 in the four main nervous territories of the forearm (ulnar, median, radial, musculocutaneous) using the score described by Boivin et al. after the surgery.
  A score of 0 to 2 will be assigned according to the motor response (0 = Normal force compared to the contralateral side, 1 = Decrease in force (possible movement against gravity) compared to the contralateral side, 2 = no movement possible)
Proportion of patients presenting at least a partial sensory block in the four main nervous territories of the forearm | 24 hours after surgery
  Proportion of patients presenting at least a partial sensory block in the four main nervous territories of the forearm (ulnar, median, radial and musculocutaneous) using the score described by Boivin et al. after the surgery.
  A score of 0 to 2 will be assigned for each dermatome (0 = normal feeling; 1 = reduced sensation compared to the contralateral side (hypoesthesia); 2 = no feeling (anesthesia)).
Time to complete catheter placement | Day of surgery, after catheter placement
  The time needed to complete catheter placement by the anesthesiologist in seconds
Occurrence of adverse events during the block | Day of surgery, after catheter placement
  The adverse events occurring during the block will be noted, such as vascular punctures, pneumothorax, paresthesias, repositioning for failure to raise the catheter through the needle.
Rate of complete sensory block | Day of surgery, 30 minutes after catheter placement
  Proportion of patients presenting at least a partial sensory block in the four main nervous territories of the forearm (ulnar, median, radial and musculocutaneous) using the score described by Boivin et al., 30 minutes after the catheter placement.
  A score of 0 to 2 will be assigned for each dermatome (0 = normal feeling; 1 = reduced sensation compared to the contralateral side (hypoesthesia); 2 = no feeling (anesthesia)).
Rate of complete motor block | Day of surgery, 30 minutes after catheter placement
  Proportion of patients presenting a motor block score greater than or equal to 1 in the four main nervous territories of the forearm (ulnar, median, radial, musculocutaneous) using the score described by Boivin et al., 30 minutes after the catheter placement.
  A score of 0 to 2 will be assigned according to the motor response (0 = Normal force compared to the contralateral side, 1 = Decrease in force (possible movement against gravity) compared to the contralateral side, 2 = no movement possible)
Worst pain during the block technique | Day of surgery, after catheter placement
  Worst pain during the block technique assessed using a numerical scale where 0 = no pain and 10 = worst pain imaginable.
Total opioid consumption | 24 and 48 hours after surgery
Time between the end of surgery and the first opioid dose | 24 hours after surgery
Minimum pain after the surgery | 24 and 48 hours after surgery
  Minimum pain reported by the patient, rated on a numerical scale where 0 = no pain and 10 = worst pain imaginable.
Maximum pain after the surgery | 24 and 48 hours after surgery
  Maximum pain reported by the patient, rated on a numerical scale where 0 = no pain and 10 = worst pain imaginable.
Average pain after the surgery | 24 and 48 hours after surgery
  Average pain reported by the patient, rated on a numerical scale where 0 = no pain and 10 = worst pain imaginable.
Percentage of time spent with moderate to severe pain | 24 and 48 hours after surgery
  Percentage of time spent with moderate to severe pain (> 4/10) using a numerical scale where 0 = no pain and 10 = worst pain imaginable
Rate of complications or adverse effects | 48 hours after surgery
  The rate of complications or adverse effects during the first 48 hours will be assessed, such as local anesthetic toxicity, nausea, vomiting, dizziness, drowsiness and accidental withdrawal of the catheter.
Quality of sleep | 24 hours and 48 hours after surgery
  The quality of sleep of the patient will be evaluated, rated on a scale where 0 = insomnia and 10 = excellent quality sleep.
Patient's satisfaction | 48 hours after surgery
  The satisfaction of the patient will be evaluated, rated on a scale where 0 = completely dissatisfied and 10 = fully satisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Maxim Roy, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada